CLINICAL TRIAL: NCT00851773
Title: A Randomised, Double Blind, Placebo-controlled, Parallel-group, Multiple Doses, Dose Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics Profiles of NN9535 in Healthy Male Japanese and Caucasian Subjects After Weekly Subcutaneous Injections.
Brief Title: Safety, Tolerability, and Profile of Action of Drug in the Body of NN9535 in Healthy Male Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-3633; 2008-006325-13 (EudraCT Number)
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- A (Experimental)
  Interventions: Drug: semaglutide
- B (Experimental)
  Interventions: Drug: semaglutide
- C (Experimental)
  Interventions: Drug: semaglutide
- D (Experimental)
  Interventions: Drug: semaglutide
- E (Experimental)
  Interventions: Drug: semaglutide
- F1 (Placebo Comparator)
  Interventions: Drug: placebo
- F2 (Placebo Comparator)
  Interventions: Drug: placebo
- F3 (Placebo Comparator)
  Interventions: Drug: placebo
- F4 (Placebo Comparator)
  Interventions: Drug: placebo
- F5 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: semaglutide — 0.1 mg once weekly, s.c. injection
  Arms: A
Drug: semaglutide — 0.2 mg once weekly, s.c. injection
  Arms: B
Drug: semaglutide — 0.4 mg once weekly, s.c. injection
  Arms: C
Drug: semaglutide — 0.4 mg once weekly for 1 week, 0.8 mg once weekly for 7 weeks, s.c. injection
  Arms: D
Drug: semaglutide — 0.4 mg once weekly for 1 week, 0.8 mg once weekly for 1 week, 1.2 mg once weekly for 6 weeks, s.c. injection
  Other Names: NN9535
  Arms: E
Drug: placebo — 0.1 mg once weekly, s.c. injection
  Arms: F1
Drug: placebo — 0.2 mg once weekly, s.c. injection
  Arms: F2
Drug: placebo — 0.4 mg once weekly, s.c. injection
  Arms: F3
Drug: placebo — 0.4 mg once weekly for 1 week, 0.8 mg once weekly for 7 weeks, s.c. injection
  Arms: F4
Drug: placebo — 0.4 mg once weekly for 1 week, 0.8 mg once weekly for 1 week, followed by 1.2 mg once weekly injections for 6 weeks, s.c. injection
  Arms: F5

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to assess and compare the safety and tolerability, as assessed by adverse events after multiple subcutaneous doses of NN9535 in healthy male Japanese and Caucasian subjects.

ELIGIBILITY:
Inclusion Criteria:

* For Caucasian or Japanese volunteers the following applies:
* Informed consent obtained before any trial-related activities
* Body weight between 54 and 90 kg (both inclusive)
* Body mass index (BMI) between 18.5 and 24.9 kg/m2 (both inclusive)
* HbA1c below 6.0 %
* Subjects who are considered to be generally healthy based on assessment of medical history, physical examination and clinical laboratory data at screening, as judged by the Investigator
* Subjects who are sexually active and have partners who are or could be pregnant are willing and required to use a barrier method of contraception (e.g. condom) for the duration of the study and for 90 days following the last dose of study medication
* Japanese passport holder, Japanese-born parents, lived outside Japan for 5 years or less

Exclusion Criteria:

* Any clinical laboratory values deviating from or outside the laboratory reference range unless considered not to be clinically significant by the investigator
* Any abnormal ECG findings at the screening, considered to be clinically significant by the Investigator
* Presence or history of diabetes, cancer or any clinically significant cardiac, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, dermatological, venereal, haematological, neurological, or psychiatric diseases or disorders, considered to be clinically significant by the Investigator
* Previous randomised in this trial (not applicable for stand-by volunteers)
* Blood pressure in supine position at the screening, after resting for 5 min, and in the standing position after standing for 1 min, consistently outside the ranges 90 - 140 mmHg systolic or 40 - 90 mmHg diastolic
* Heart rate in supine position at the screening, after resting for 5 min, consistently above 100 beats/min
* Alcohol intake within 48 hours prior to the screening and admission (examined by alcohol breath test)
* Hepatitis B surface antigen, Hepatitis C antibodies or Human Immunodeficiency Virus (HIV) antibodies positive
* History of significant allergy or hypersensitivity
* Known or suspected allergy to trial product or related products
* History of drug or alcohol abuse (alcohol abuse is defined as intake of more than 21 units (U) weekly: One unit of alcohol equals 1/2 pint (approximately 250 mL) of beer or lager, or one glass of wine or Japanese sake, or 1/6 gill (approximately 20 mL) of spirits)
* Subjects who smoke more than 10 cigarettes, or the equivalent, per day or is unwilling to refrain from smoking whenever required for the trial procedure
* Use of prescription drugs within 3 weeks prior to dosing, non-prescription drugs within 1 week prior to dosing except for vitamins, minerals and nutritional supplements
* Received any investigational drug within 12 weeks prior to the planned first dosing
* Subjects who have taken part in strenuous exercise within 48 hours prior to first dosing, due to interference with the hepatic microsomal monooxygenase system. The Investigator or Sub-Investigator will evaluate whether strenuous exercise has been undertaken
* Loss of more than 400 mL blood in total within the last 12 weeks or more than 200 mL blood in total within the last 4 weeks prior to first dosing
* Subjects with a first-degree relative with diabetes mellitus
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Possibility that the subject will not comply with the protocol
* Subjects who in the opinion of the Investigator or Sub-Investigator should not participate in the trial
* Subjects with known history of either Type 1 or Type 2 diabetes mellitus are excluded

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Adverse events | at all scheduled visits (2 - 14) following screening

SECONDARY OUTCOMES:
Frequency of hypoglycaemic episodes | at all scheduled visits (2 - 14) following screening
Vital signs (blood pressure and pulse) | at all scheduled visits (2 - 14) including screening (visit 1)
12-lead ECG (electrocardiogram) | at all scheduled visits (2 - 14) including screening (visit 1)
Haematology | at all scheduled visits (2 - 14) including screening (visit 1)
Biochemistry | at all scheduled visits (2 - 14) including screening (visit 1)
Urinalysis | at all scheduled visits (2 - 14) including screening (visit 1)
Calcitonin | at screening (visit 1) and at visits 2, 9 and 14
Antibody development against N9535 | at visits 2 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- London Southwest, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com